CLINICAL TRIAL: NCT04150159
Title: Evaluation of a Fasting Mimicking Diet and the Effect on Endothelial Function, Body Composition and Vascular Markers
Brief Title: Evaluation of a Fasting Mimicking Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hypertension Institute, Nashville (Other)
Collaborators: L-Nutra Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HTI 001
Record Dates: First submitted 2019-10-25; First posted 2019-11-04 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: This is a randomized, open-label, 7-month trial in eighty (80) adult subjects. Forty (40) subjects will be randomized to the intervention FMD arm with a 5 day meal program every month for four (4) months. Forty subjects will be randomized to a follow a Mediterranean diet plan for four months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting Mimicking Diet (FMD) Arm (Experimental): The ProLon® FMD diet is made up of nut bars, dehydrated soups, tea, olives, kale crackers, electrolyte beverages, and a chocolate crisp bar consumed for 5 days every 30 days for 4 months.
  Interventions: Dietary Supplement: FMD Arm
- Mediterranean Diet Arm (Active Comparator): The Mediterranean diet is based on the traditional foods that people used to eat in countries like Italy and Greece in the 1960s.
  * Eat every day: vegetables, fruits, nuts, seeds, legumes, potatoes, whole grains, breads, yogurt, dairy, fish/seafood, herbs, spices and extra virgin olive oil.
  * Eat three or fewer servings each week: poultry, eggs, cheese.
  * Eat two or fewer servings each week: red meat, potatoes.
  * Eat two or fewer servings each week: sweets, sodas, processed meat, refined grains, refined oils and other highly processed foods.
  Interventions: Dietary Supplement: FMD Arm

INTERVENTIONS:
Dietary Supplement: FMD Arm — ProLon Fasting Mimicking Diet Plan

SUMMARY:
Randomized, open-label, 7-month trial in eighty (80) adult subjects. Forty (40) subjects will be randomized to the intervention FMD arm with a 5 day meal program every month for four (4) months. Forty subjects will be randomized to a follow a Mediterranean diet plan for four months. Both arms will have a final study visit at month 7.

DETAILED DESCRIPTION:
Determine the effects of the FMD on cardiovascular (CV) biomarkers, coronary heart disease (CHD) risk factors (body weight, body mass index (BMI), body composition, blood pressure, serum lipid levels and dysglycemia blood measurements), noninvasive cardiovascular testing for endothelial function, arterial stiffness of large and small arteries and autonomic function testing in adult subjects over a seven-month study period.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index equal to or greater than 28
* EndoPAT® Score for endothelial function of less than or equal to 2.0 or AC 2 small resistance artery compliance by computerized arterial pulse wave analysis (CAPWA) of less than or equal to 5.0.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Individuals who are allergic to tree nuts (macadamia, cashew, almond, pecan), soy, oats, sesame, or celery/celeriac
* Pregnant females
* Any cancer within the past 5 years
* Documented myocardial infarction within past 5 years
* Documented cerebrovascular accident within past 5 years
* Chronic steroid use (longer than 45 consecutive days
* Type I insulin-dependent diabetes mellitus

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to End of Study in endothelial function | 7 months
  Endothelial function will be measured for all subjects with EndoPAT and PulseWave noninvasive testing and laboratory analysis markers

SECONDARY OUTCOMES:
Change from Baseline to End of Study in cardiovascular biomarkers | 7 months
  Cardiovascular biomarkers will be measured for all subjects with serum lipid levels and serum inflammatory markers

CONTACTS AND LOCATIONS:
Locations (1):
- Hypertension Institute, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No